CLINICAL TRIAL: NCT00471211
Title: A 12-Week, Randomised, Double-Blind, Placebo-Controlled, Parallel Three-Group Study to Assess the Safety, Tolerability and Efficacy of Two Dose Levels of PBT2 to Slow Progression of Disease in Patients With Early Alzheimer's Disease
Brief Title: Study Evaluating the Safety, Tolerability and Efficacy of PBT2 in Patients With Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prana Biotechnology Limited (Industry)
Organization: Pranabio (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBT2-201
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PBT2

SUMMARY:
The purpose of the study is to determine the safety, tolerability and efficacy of 2 doses of PBT2 administered for 12 weeks compared to placebo in patients with early Alzheimer's disease treated with an acetylcholinesterase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of probable early Alzheimer's disease
* stable dose of acetylcholinesterase inhibitor
* community dwelling
* stable medical condition

Exclusion Criteria:

* unstable and significant medical conditions
* recurrent major psychiatric disorder
* treatment with memantine

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety | Study duration

SECONDARY OUTCOMES:
Change from baseline in biomarkers; Change from baseline in cognitive and global function scales | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lannfelt, Professor, Principal Investigator — Uppsala University Hospital, Sweden
Locations (11):
- Australia (3):
  - Sydney, New South Wales
  - Adelaide, South Australia
  - Melbourne, Victoria
- Sweden (8):
  - Falköping
  - Kalix
  - Kalmar
  - Lund
  - Malmo
  - Stockholm
  - Umeå
  - Uppsala

REFERENCES:
- [Derived] Lannfelt L, Blennow K, Zetterberg H, Batsman S, Ames D, Harrison J, Masters CL, Targum S, Bush AI, Murdoch R, Wilson J, Ritchie CW; PBT2-201-EURO study group. Safety, efficacy, and biomarker findings of PBT2 in targeting Abeta as a modifying therapy for Alzheimer's disease: a phase IIa, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2008 Sep;7(9):779-86. doi: 10.1016/S1474-4422(08)70167-4. Epub 2008 Jul 30. PMID 18672400